CLINICAL TRIAL: NCT05588024
Title: International Device Assisted Controlled Sequential Elevation CPR Registry
Status: Recruiting | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Johanna Moore, Johanna Moore, MD MSc, Hennepin Healthcare Research Institute
Other Study IDs: 1281037
Record Dates: First submitted 2022-07-01; First posted 2022-10-20 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Arrest, Out-Of-Hospital
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Head Up CPR based bundle of care: All patients in the registry receive the Head Up CPR based bundle of care.
  Interventions: Device: Head Up CPR based bundle of care

INTERVENTIONS:
Device: Head Up CPR based bundle of care — All patients in this registry receive the intervention, a Head Up Cardiopulmonary Resuscitation (CPR) based bundle of care. This bundle of care includes the use of multiple FDA approved devices. The components of the Head Up CPR bundle are 1) a single or combination of CPR methods including manual, active-compression decompression CPR, or automated suction-cup based CPR 2) An impedance threshold device 3) An automated patient positioning device capable of elevating the head and thorax

SUMMARY:
The purpose of this prospective observational cardiopulmonary resuscitation (CPR) registry is to track the use and clinical outcomes from emergency medical systems across the US and Europe that have implemented a system of care approach applied rapidly to cardiac arrest that includes using the combination of an impedance threshold device (ITD), and either manual active compression-decompression (ACD) CPR device or automated compression device, with a Head Up CPR device.

DETAILED DESCRIPTION:
In 2019, a FDA approved patient positioning device capable of elevating the head and thorax in a controlled manner became commercially available. As emergency medical services are increasingly using this Head Up CPR patient positioning device as part of their standard protocol for cardiac arrest patients, in addition to Active Compression-Decompression (ACD) cardiopulmonary resuscitation with an Impedance Threshold Device (ITD) CPR or with mechanical CPR and the ITD, it is important to monitor how this device is being used, and outcomes of patients who received this Head Up CPR therapy. All of the devices used in this observational registry study have received FDA 510K clearance.

Emergency medical systems (EMS) that have implemented standard cardiac arrest protocols that include the combination of manual CPR with an ITD, an automated CPR device with the ITD, or ACD+ITD CPR, with the Head Up CPR device are asked to be part of the Registry. If a system participates, they are asked for de-identified cardiac arrest data including patient demographics, details of cardiac arrest care, and patient outcomes before and after implementation of the Head Up CPR bundle. De-identified data is kept securely by the study sponsor and PI. The patient data for all systems using this approach to resuscitation are included, with a current focus on patients receiving the device combination rapidly.

ELIGIBILITY:
Inclusion Criteria

1. Patient is at least 18 years of age
2. Patient is in active cardiac arrest, as defined by presence of either ventricular fibrillation or ventricular tachycardia, or pulseless electrical activity, or asystole at time of enrollment.
3. Patient receives either a) active-compression decompression cardiopulmonary resuscitation b) automated suction-cup based CPR with an impedance threshold device (ITD) c) manual CPR with an ITD
4. Subject receives device assisted controlled elevation of the head and thorax.

Exclusion Criteria

1. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with out-of-hospital cardiac arrest in areas where emergency medical services that have a Head Up CPR based system of care in their cardiac arrest protocol as part of routine clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-03-23 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Return of Spontaneous Circulation | From the start of CPR to the presence of cardiac activity. The time period in which this outcome will varies and is estimated to range from 0 minutes up to around 40 minutes.
  Presence of cardiac activity with a perfusing blood pressure
Survival | The time period in which this outcome will occur will vary, may extend up to 60 days.
  If the patient survived admission to the hospital until hospital discharge
Survival with Favorable Neurological Function | The time period in which this outcome will occur will vary, may extend up to 60 days.
  If the patient survived admission to the hospital until hospital discharge with favorable Cerebral Performance Category (CPC) Score as defined CPC 1 or 2.

SECONDARY OUTCOMES:
End tidal CO2 (ETCO2) | ETCO2 will be measured continuously while the patient is receiving CPR. This time period is estimated to occur up to 40 minutes.
  ETCO2 is an indirect measure of perfusion during CPR
Cerebral Oximetry | If the participating EMS system in the registry uses NIRS cerebral oximetry, it will be measured continuously while the patient is receiving CPR. This time period is estimated to occur up to 40 minutes.
  Near-infrared spectroscopy (NIRS) capable of measuring regional tissue oxygenation.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna C Moore, MD, MS, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin Healthcare Research Institute, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore JC, Pepe PE, Scheppke KA, Lick C, Duval S, Holley J, Salverda B, Jacobs M, Nystrom P, Quinn R, Adams PJ, Hutchison M, Mason C, Martinez E, Mason S, Clift A, Antevy PM, Coyle C, Grizzard E, Garay S, Crowe RP, Lurie KG, Debaty GP, Labarere J. Head and thorax elevation during cardiopulmonary resuscitation using circulatory adjuncts is associated with improved survival. Resuscitation. 2022 Oct;179:9-17. doi: 10.1016/j.resuscitation.2022.07.039. Epub 2022 Aug 4. PMID 35933057
- [Background] Bachista KM, Moore JC, Labarere J, Crowe RP, Emanuelson LD, Lick CJ, Debaty GP, Holley JE, Quinn RP, Scheppke KA, Pepe PE. Survival for Nonshockable Cardiac Arrests Treated With Noninvasive Circulatory Adjuncts and Head/Thorax Elevation. Crit Care Med. 2024 Feb 1;52(2):170-181. doi: 10.1097/CCM.0000000000006055. Epub 2024 Jan 19. PMID 38240504
- [Background] Moore JC, Duval S, Lick C, Holley J, Scheppke KA, Salverda B, Rojas-Salvador C, Jacobs M, Nystrom P, Quinn R, Adams PJ, Debaty GP, Hutchison M, Mason C, Martinez E, Mason S, Clift A, Antevy P, Coyle C, Grizzard E, Garay S, Lurie KG, Pepe PE. Faster time to automated elevation of the head and thorax during cardiopulmonary resuscitation increases the probability of return of spontaneous circulation. Resuscitation. 2022 Jan;170:63-69. doi: 10.1016/j.resuscitation.2021.11.008. Epub 2021 Nov 15. PMID 34793874